CLINICAL TRIAL: NCT04417452
Title: Effects of Fetal Programming on the Metabolic, Cardiovascular, Neurocognitive and Reproductive Health of Offsprings and Their Mothers After Pregnancies With Diabetes
Brief Title: Long-term Outcome After Gestational Diabetes and Diabetes in Pregnancy
Acronym: MuKiLOG
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Jena University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-1403
Record Dates: First submitted 2020-04-15; First posted 2020-06-04 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Diabetes, Gestational; Pregnancy Diabetic
MeSH Terms: conditions — Diabetes, Gestational | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mothers / children after diabetes in pregnancy: The study collective is composed of mother-child pairs after gestational diabetes, which were supervised in the Competence Center for Diabetes and Pregnancy at the University Hospital of Jena. The patients can decide to fill in an online questionnaire. For all other parts of the study, only patients who have been informed individually or on behalf of their legal guardian about the nature of the study after a detailed and understandable explanatory discussion with an investigator and who have given written consent will be included in the study.
  Interventions: Other: Basic data collection (online survey or written form); Other: Physical examination; Behavioral: Psychometric examination; Diagnostic Test: Recording of the adrenergic stress reaction (saliva test)
- Controls: The control collective is composed of mother-child pairs who were cared for at the same time as the study collective at the University Hospital Jena. This collective is status post singleton pregnancy and term birth. The patients can decide to fill in an online questionnaire. For all other parts of the study, only patients who have been informed individually or on behalf of their legal guardian about the nature of the study after a detailed and understandable explanatory discussion with an investigator and who have given written consent will be included in the study.
  Interventions: Other: Basic data collection (online survey or written form); Other: Physical examination; Behavioral: Psychometric examination; Diagnostic Test: Recording of the adrenergic stress reaction (saliva test)

INTERVENTIONS:
Other: Basic data collection (online survey or written form) — Basic data collection is carried out by means of a questionnaire that participants can fill in outside the study centre. It contains questions about the current life situation, sleep and activity behaviour.
Other: Physical examination — The physical examination takes place at the study centre and includes the measurement of height, current weight and body fat, as well as the recording of heart and circulation parameters (e.g. blood pressure measurement or determination of vascular health by means of ultrasound). General metabolic and hormonal parameters are analysed by means of a blood sample. In addition, a sugar test for diabetes diagnosis will be carried out.
Behavioral: Psychometric examination — Psychometric examination is carried out at the study centre with the help of a RIAS (Reynolds Intellectual Assessment Scales and Screening) test.
Diagnostic Test: Recording of the adrenergic stress reaction (saliva test) — The adrenergic stress reaction is recorded by a saliva test.

SUMMARY:
The primary objectives of the proposed project are to assess the long-term effects of prenatal exposure to gestational diabetes or diabetes on the maturation and health of the offspring. In addition, the long-term changes on the health of the affected mothers will be investigated, taking into account the metabolic adjustment during index pregnancy. The expected results will help to establish possible prevention strategies to fight the epidemic of non-communicable diseases for the offspring and the mothers.

DETAILED DESCRIPTION:
Investigation of the long-term outcome of mother-child pairs after diabetic pregnancies and a comparison group regarding metabolic, cardiovascular, neurocognitive and reproductive long-term changes as a function of the course of pregnancy and metabolic control

ELIGIBILITY:
Inclusion Criteria:

* For the pilot project: Initial participation in the preliminary study
* Written Informed Consent
* Singleton pregnancies
* Delivery at the University Hospital Jena

Exclusion criteria:

* Severe physical and mental illness
* Patients who refuse to participate in the study or drop out
* Premature birth, i.e. birth of the child <37/0 weeks of gestation
* Serious pregnancy complications
* Prenatally known serious malformations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study collective is composed of mother-child pairs after gestational diabetes, which were supervised in the Competence Center for Diabetes and Pregnancy at the University Hospital of Jena. The patients can decide to fill in an online questionnaire. For all other parts of the study, only patients who have been informed independently or on behalf of their legal guardian about the nature of the study after a detailed and understandable explanatory discussion with an investigator and who have given written consent will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Metabolic health | 1 day examination at the study centre
  effects on metabolic health such as glucose tolerance disorders and diabetes mellitus, obesity and metabolic syndrome (mothers and children)
Neurocognitive development | 1 day examination at the study centre
  effects on neurocognitive development, mental health and adrenal and autonomic stress reactivity (mothers and children)
Cardiovascular and vascular health | 1 day examination at the study centre
  effects on cardiovascular and vascular health of blood pressure regulation and endothelial function (mothers and children)
Maturation of the gonadal regulation | 1 day examination at the study centre
  maturation of gonadal regulation, pubertal development and reproductive health (children)

CONTACTS AND LOCATIONS:
Overall Officials: Friederike Weschenfelder, Dr. med., Principal Investigator — Klinik für Geburtsmedizin
Locations (1):
- Universitätsklinikum Jena, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No